CLINICAL TRIAL: NCT05530993
Title: Exploring the Perspectives and Experiences of PrEP-eligible Black Women in Texas in Relation to Readiness for PrEP Uptake and Adherence
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mandy Hill, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-22-0565
Record Dates: First submitted 2022-08-25; First posted 2022-09-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: PrEP Uptake Perspectives; PrEP Uptake Experiences; PrEP Adherence Perspectives; PrEP Adherence Experiences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Have considered use of PrEP
- Have not considered use of PrEP

SUMMARY:
The aim is to conduct two virtual focus groups (10 participants in each group) with 20 pre-exposure prophylaxis (PrEP)-eligible Black women in Houston and Austin, TX. Participants will be assigned to focus groups with other women based on their position about PrEP uptake (considered use versus not considered use). Focus group questions will build on an ecologic model framework to inquire about participant's intrapersonal, interpersonal, and community-level factors that influence access to and use of HIV prevention services. This strategy aims to examine potential barriers to PrEP uptake among PrEP-eligible women in two Texas' hotspots.

ELIGIBILITY:
Inclusion Criteria:

* assigned female sex at birth
* identify as Black or African American
* 18 years of age or older
* have had condomless sex with a cisgender man within the past 12 months
* fluent in English or Spanish
* have a phone or internet access
* not currently on PrEP and have never taken PrEP

Exclusion Criteria:

* choose not to identify as Black or African American
* unable to provide informed consent for participation (e.g. have severe cognitive impairment that would interfere with their ability to consent)
* have psychological distress that would prohibit them from participating in the study
* unable or unwilling to meet study requirements
* ineligible for HIV prevention services [i.e., Human Immunodeficiency Virus (HIV) Positive]
* received a prescription for PrEP within 12 months
* has a history of PrEP uptake or is currently on PrEP

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as a woman.
Study Population: PrEP-eligible Black women in Harris County of Houston, TX and Travis County of Austin, TX will be recruited. An e-flyer will be distributed through the social media networks of academic and community partners, with potential for sharing amongst their followers to their social media following.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Facilitators to readiness to adopt PrEP | during the focus group
  A focus group will be used to identify facilitators to readiness to adopt PrEP (a focus group is a group interview among the study participants with the purpose of collecting information about a topic, in this case facilitators to readiness to adopt PrEP). During the focus group, focus group participants will be asked to indicate facilitators to readiness to adopt PrEP, and these facilitators to readiness will be recorded at the time of the focus group. These facilitators to readiness identified during the focus group will be reported categorically.
Barriers to readiness to adopt PrEP | during the focus group
  A focus group will be used to identify barriers to readiness to adopt PrEP (a focus group is a group interview among the study participants with the purpose of collecting information about a topic, in this case barriers to readiness to adopt PrEP). During the focus group, focus group participants will be asked to indicate barriers to readiness to adopt PrEP, and these barriers to readiness will be recorded at the time of the focus group. These barriers to readiness identified during the focus group will be reported categorically.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy J Hill, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - The University of Texas at Austin, Austin, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No